CLINICAL TRIAL: NCT02513082
Title: Effectiveness of Pain Relief Between Adductor Canal Block and Femoral Nerve Block in Total Knee Arthroplasty in General Anesthesia
Brief Title: Effectiveness of Pain Relief Between Adductor Canal Block and Femoral Nerve Block in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nerve block
Record Dates: First submitted 2015-07-28; First posted 2015-07-31 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femoral nerve block (Experimental): Femoral nerve block will be performed just one time after total knee arthroplasty in general anesthesia state
  Interventions: Procedure: Sono guided nerve block
- Adductor canal block (Active Comparator): Adductor canal block will be performed just one time after total knee arthroplasty in general anesthesia state
  Interventions: Procedure: Sono guided nerve block

INTERVENTIONS:
Procedure: Sono guided nerve block — Sono guided nerve block is effectively and safely performed for pain relief after total knee arthroplasty
  Other Names: femoral nerve block; adductor canal block

SUMMARY:
This study aims to compare the effectiveness of adductor canal block and femoral nerve block in total knee arthroplasty in general anesthesia. Two block techniques were proved safe and effective in pain control after total knee arthroplasty. But some authors insist that quadriceps muscle power was decreased by femoral nerve block. The study design is a double-blind randomized controlled trial. Fifty patients planed to undergo simultaneously bilateral total knee arthroplasty are randomised to receive ultrasound-guided femoral nerve block on one leg and adductor canal block on the other, in addition to combined general anaesthesia. The primary outcome was comparative postoperative pain in either extremity at four, eight, 12, 24, 72 hours and 7days postoperatively. Secondary comparative outcomes included motor strength by cybex test.

DETAILED DESCRIPTION:
Total knee arthroplasty(TKA) is very popular in nowadays. But almost patients complained of postoperative pain and it affect the delay of early mobilization which prevent knee stiffness, lessens hospital stay and improves overall patient satisfaction and outcome of TKA. Intravenous patient-controlled analgesia (PCA) or epidural analgesia is a conventional postoperative analgesia. Recently other block techniques like a adductor canal block and femoral nerve block were known for good methods of pain relief after TKA. However, femoral nerve block reduces quadriceps muscle strength thereby potentially compromising postoperative mobilization. Therefore, it is necessary to evaluate the effectiveness of pain treatment and the preservation of muscle function after the procedure of adductor canal block and femoral nerve block.

The present study aimed to determine and compare the efficacy of adductor canal block and femoral nerve block combined with general anesthesia on (1) postoperative pain control, (2) early patient ambulation and functional recovery and (3) change of muscle power after total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients for total knee arthroplasty having medicare insurance

Exclusion Criteria:

* Alcohol, drug abuser Narcotics addiction

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Changes in Visual pain scale | Changes from the baseline visual pain scale to 1 week after surgery

SECONDARY OUTCOMES:
Changes in Quadriceps muscle power and strength by cybex muscle testing | 1 week postoperatively compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yong In, MD, PhD, Study Chair — the Catholic Univerisity of Korea Seoul St Mary's hospital

REFERENCES:
- [Derived] Koh HJ, Koh IJ, Kim MS, Choi KY, Jo HU, In Y. Does Patient Perception Differ Following Adductor Canal Block and Femoral Nerve Block in Total Knee Arthroplasty? A Simultaneous Bilateral Randomized Study. J Arthroplasty. 2017 Jun;32(6):1856-1861. doi: 10.1016/j.arth.2017.01.025. Epub 2017 Jan 26. PMID 28215966